CLINICAL TRIAL: NCT06636227
Title: Optimal Dosing, Tolerability, and Initial Efficacy of Diclofenac as a KMO Inhibitor in Individuals With Alcohol Use Disorder
Brief Title: Diclofenac Dose Response Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Daniel Roche, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00109891
Record Dates: First submitted 2024-10-03; First posted 2024-10-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder (AUD); Alcohol-Related Disorders
Keywords: Alcohol use disorder (AUD); Alcohol-Related Disorders; Alcoholism; Drinking Behavior; Substance-Related Disorders; Chemically-Induced Disorders
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders; Drinking Behavior; Substance-Related Disorders; Chemically-Induced Disorders | interventions — Diclofenac

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled, randomized, cross-over study in which individuals with AUD (n=24) complete four sessions where they receive diclofenac (50 mg, 75 mg, or 100 mg) or placebo. Eligible participants will be randomized to receive the three doses of diclofenac and placebo in a randomized, double-blind fashion. Because the study is completely within subject, there are no groups or group assignment. There are no control subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo control
- Diclofenac 50mg (Active Comparator): In this arm participants will receive 50mg of Diclofenac
  Interventions: Drug: Diclofenac 50mg
- Diclofenac 75mg (Active Comparator): In this arm participants will receive 75mg of Diclofenac
  Interventions: Drug: Diclofenac 75mg
- Diclofenac 100mg (Active Comparator): In this arm participants will receive 100mg of Diclofenac
  Interventions: Drug: Diclofenac 100mg

INTERVENTIONS:
Drug: Diclofenac 100mg — Diclofenac 100mg
  Arms: Diclofenac 100mg
Drug: Diclofenac 75mg — Diclofenac 75mg
  Arms: Diclofenac 75mg
Drug: Diclofenac 50mg — Diclofenac 50mg
  Arms: Diclofenac 50mg
Drug: Placebo control — Placebo control
  Arms: Placebo

SUMMARY:
The development of efficacious medications for AUD remains a high research priority with current emphases on identifying novel molecular targets and efficiently screening new compounds. Pharmacological modulation of the kynurenine pathway (KP) represents a promising novel target for AUD. The KP is a complex enzymatic cascade with each step producing biologically active metabolites that are critically involved in diverse physiological and pathological processes. Chronic alcohol exposure produces dysregulation of the KP, particularly as evidenced by decreased levels of the neuroprotective metabolite kynurenic acid (KYNA) and increased levels of the neurotoxic metabolite quinolinic acid (QUIN). This metabolic shift is associated with various alcohol-related pathologies in animals and humans. Thus, a medication that targets the KP to restore KYNA and attenuate QUIN levels may be an effective treatment for AUD. The enzyme kynurenine 3- monooxygenase (KMO) is a major gatekeeper of the KP and resultant KYNA levels. KMO inhibition shifts the KP towards KYNA production in brain and away from QUIN production. Critically, KMO inhibition in rodents, through its increase in brain KYNA levels, decreases alcohol self-administration, preference, cue-reactivity, and relapse behaviors. However, KMO-inhibitors have not been tested in humans because of presumed lack of availability. Diclofenac is an FDA-approved Non-Steroidal Anti-Inflammatory Drug that was recently discovered to inhibit KMO activity. Consistent with KMO inhibition, diclofenac increases KYNA levels in the brain and periphery of rodents. However, it remains unknown whether diclofenac increases KYNA levels and affects alcohol-related behaviors in humans at approved, safe dosages.

Investigators propose to conduct a human laboratory pilot study to test whether diclofenac can increase KYNA in individuals with AUD, and if so, which of 3 doses (50, 75, or 100 mg) most effectively increases KYNA. Individuals with AUD (n = 24) will complete four sessions where they receive diclofenac (50, 75, or 100 mg) or placebo. Investigators will examine increases in KYA levels and will also assess QUIN levels, alcohol craving, and negative mood.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is a chronic condition for which current pharmacological treatments are only modestly effective [1,2]. The development of efficacious medications for AUD remains a high research priority with current emphases on identifying novel molecular targets and efficiently screening new compounds for AUD [3,4]. To that end, modulation of the kynurenine pathway (KP) represents a promising novel target for AUD.

The KP is a complex enzymatic cascade with each step producing biologically active metabolites that are critically involved in diverse physiological and pathological processes. Accumulating evidence suggests that chronic alcohol exposure produces dysregulation of the KP, particularly as evidenced by altered levels of the metabolites kynurenic acid (KYNA) and quinolinic acid (QUIN). KYNA is an NMDA receptor and α7 nicotinic acetylcholine receptor (nAChR) antagonist that has neuroprotective and anticonvulsant properties [5,6]. Conversely, QUIN is an NMDA receptor agonist containing neurotoxic and convulsant properties [7-9]. Both NMDA and α7nAChR are critically involved in addiction neurobiology. For example, α7nAChRs control glutamate release from cortical afferents to the nucleus accumbens and thereby modulate mesolimbic dopamine release in response to acute alcohol consumption and alcohol-related cues [10-12]. Chronic alcohol exposure produces ametabolic shift away from KYNA and toward QUIN production, and this imbalance is associated with various alcohol-related pathologies in animals and humans [11-14]. Thus, a medication that targets the KP to restore KYNA and attenuate QUIN levels may hold promise as an effective treatment for AUD.

The enzyme kynurenine 3-monooxygenase (KMO) is increasingly understood to be a major gatekeeper of the KP and its production of KYNA. KMO inhibition shifts the KP towards KYNA production in the brain [15], whereas KMO upregulation shifts the KP toward QUIN production. Critically, KMO inhibition in rodents decreases alcohol self-administration, alcohol preference, relapse to alcohol consumption, and cue-induced reinstatement of alcohol-seeking [11,12,16]. These anti-alcohol effects were predominantly due to brain increases in KYNA, which blocked alcohol-induced dopamine release in the nucleus accumbens shell through antagonism of α7nAChreceptors11,12. KMO inhibition also reduced nicotine- and cannabinoid-induced extracellular dopamine release in the nucleus accumbens shell, self-administration of nicotine and cannabinoids, cue-induced nicotine and cannabinoid relapse behaviors, and cocaine-seeking behavior; like with alcohol, these effects were also in part to KYNA's antagonism of α7nACh receptors [11,17-19]. These preclinical findings suggest increasing KYNA levels though KMO inhibition is a promising target for the treatment of AUD as well as other substances of misuse, but medications with this pharmacological property have not been tested in humans.

Diclofenac is an FDA-approved Non-Steroidal Anti-Inflammatory Drug (NSAID), and like all NSAIDs produces anti-inflammatory, antipyretic, and analgesic effects at least in part through inhibiting prostaglandin activity. However, it was recently discovered that diclofenac also potently inhibits KMO activity and that it may be the only FDA-approved medication with this pharmacological property [20,21]. Consistent with KMO inhibition, diclofenac increases KYNA levels in the brain and peripheral tissue in rodents [22,23]. Thus, diclofenac has a unique and promising pharmacological profile for AUD treatment. However, it remains unknown whether diclofenac increases KYNA levels in humans at approved, safe dosages, and if KMO inhibition in humans is a viable pharmacological target for treating AUD. As diclofenac is currently available and used by millions of patients each year for other indications, the repurposing of diclofenac for the treatment of AUD represents a fast and economically feasible approach to drug development.

The first step in determining whether diclofenac can be repurposed for AUD is to determine whether the drug inhibits KMO at FDA-approved safe and tolerable doses. Thus, investigators propose to conduct a human laboratory pilot study to test whether diclofenac can increase KYNA in individuals with AUD. An increase in KYNA would support the proposed pharmacological property of KMO inhibition. Individuals with AUD (n = 24) will complete four sessions where they receive one of three doses of diclofenac (50, 75, or 100 mg) or placebo. Investigators will examine increases in KYA levels and will also assess QUIN levels, alcohol craving, and negative mood.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65
* Meet DSM-5 diagnostic criteria for current AUD of any severity (Mild, Moderate, or Severe)
* In the 30-day period before enrollment, consume > 14 and > 7 standard drinks per week for men and women, respectively
* In the 30-day period before enrollment, engage in heavy drinking (5 or more drinks for men, 4 or more drinks for women) ≥ 5 times per month

Exclusion Criteria:

* Currently in treatment, a history of treatment within the 30 days before enrollment, or currently seeking immediate treatment for AUD
* Current (last 12 months) DSM-5 diagnosis of SUD for any psychoactive substances other than alcohol, nicotine, and cannabis (cannabis use disorder, mild severity allowed; moderate and severe excluded)
* Currently prescribed a psychotropic medication for the treatment of schizophrenia spectrum and other psychotic disorders, bipolar and related disorders
* Lifetime DSM-5 diagnosis of schizophrenia spectrum and other psychotic disorders and bipolar and related disorders
* Positive urine toxicology screen for the following substances: cocaine, opiates, amphetamines, methamphetamine, phencyclidine, barbiturates, benzodiazepine, methadone, and tricyclic antidepressants
* Self-reported current daily use of opioids (including prescribed)
* If female: pregnant, nursing, or with reproductive potential who refuses to use reliable methods of birth control throughout the study
* Serious alcohol withdrawal symptoms as indicated by a score ≥ 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised
* Any autoimmune disorder, inflammatory disorder, hypercoagulable state, cardiovascular disease or other medical condition (e.g., any cardiac, renal, or liver disease, uncontrolled hypertension, or diabetes) that may interfere with safe study participation and/or study aims. Specific examples of exclusionary medical conditions include but are not limited to:

  1. Any lifetime history of 1) serious GI conditions, including ulcer disease, gastrointestinal bleeding, and clinically significant gastritis, or, 2) serious cardiovascular conditions, including heart failure, myocardial infarction, stroke, pulmonary embolism, blood clots, deep vein thrombosis, or clotting disorder, 3) liver disease or impaired liver function, and 4) renal disease or insufficiency
  2. Current uncontrolled hypertension
  3. AST and ALT > four times the upper limit of the normal range, or albumin, GFR, BUN, or creatinine 15% > the upper limit of the normal range
  4. Clinically significant ECG findings, including clinically significant arrhythmia, atrioventricular block, prolonged QTc interval, or enlarged or hypertrophic heart
  5. Serious brain conditions, including epilepsy, dementia and neurodegenerative diseases, traumatic brain injury (TBI), etc. TBI exclusionary criteria include: suffered a mild or moderate TBI within the last 12 months, a severe TBI at any point in their life, or a moderate TBI before the age of 12
* Attempted suicide in the past 3 years and/or serious suicidal intention or plan within the past year
* Currently on prescription medication that contraindicates use of diclofenac, including but not necessarily limited to: oral corticosteroids, anticoagulants, lithium, warfarin, aspirin (daily use), methotrexate, cyclosporine, ACE-inhibitors, diuretics like furosemide and thiazides, and any medication that significantly influences CYP2C9 enzyme activity (e.g., rifampin, voriconazole).
* Previously known hypersensitivity, including gastroenteritis, asthma, and allergic-type reactions, to any NSAID and/or aspirin
* Current daily use of any NSAID or regular pattern of near daily use within the past three months, regular use of a prebiotic or probiotic supplement and/or any antibiotic, prebiotic, or probiotic use within the last month
* Any other circumstances that, in the opinion of the investigators, compromises participant safety, ability of the investigators to conduct the study as designed, and/or study integrity
* Current or recent (within 3 months) participation in a clinical trial involving medication administration
* Has below a 6th grade reading level
* Within the last 3 months, tested positive for COVID-19 (i.e. the SARS-CoV-2 virus) and experienced common related symptoms

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in blood kynurenic acid (KYNA) levels | From enrollment to the end of session 4 (approximately 5 weeks)
  To test whether diclofenac can increase blood kynurenic acid (KYNA) in individuals with Alcohol Use Disorder (AUD)

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rover S, Cesura AM, Huguenin P, Kettler R, Szente A. Synthesis and biochemical evaluation of N-(4-phenylthiazol-2-yl)benzenesulfonamides as high-affinity inhibitors of kynurenine 3-hydroxylase. J Med Chem. 1997 Dec 19;40(26):4378-85. doi: 10.1021/jm970467t. PMID 9435907
- [Background] Leclercq S, Schwarz M, Delzenne NM, Starkel P, de Timary P. Alterations of kynurenine pathway in alcohol use disorder and abstinence: a link with gut microbiota, peripheral inflammation and psychological symptoms. Transl Psychiatry. 2021 Oct 1;11(1):503. doi: 10.1038/s41398-021-01610-5. PMID 34599147
- [Background] Vengeliene V, Cannella N, Takahashi T, Spanagel R. Metabolic shift of the kynurenine pathway impairs alcohol and cocaine seeking and relapse. Psychopharmacology (Berl). 2016 Sep;233(18):3449-59. doi: 10.1007/s00213-016-4384-9. Epub 2016 Jul 30. PMID 27475106
- [Background] Schwarcz R, Bruno JP, Muchowski PJ, Wu HQ. Kynurenines in the mammalian brain: when physiology meets pathology. Nat Rev Neurosci. 2012 Jul;13(7):465-77. doi: 10.1038/nrn3257. PMID 22678511
- [Background] Litten RZ, Falk DE, Ryan ML, Fertig J, Leggio L. Advances in Pharmacotherapy Development: Human Clinical Studies. Handb Exp Pharmacol. 2018;248:579-613. doi: 10.1007/164_2017_79. PMID 29294197
- [Background] Maisel NC, Blodgett JC, Wilbourne PL, Humphreys K, Finney JW. Meta-analysis of naltrexone and acamprosate for treating alcohol use disorders: when are these medications most helpful? Addiction. 2013 Feb;108(2):275-93. doi: 10.1111/j.1360-0443.2012.04054.x. Epub 2012 Oct 17. PMID 23075288
- [Background] Skinner MD, Lahmek P, Pham H, Aubin HJ. Disulfiram efficacy in the treatment of alcohol dependence: a meta-analysis. PLoS One. 2014 Feb 10;9(2):e87366. doi: 10.1371/journal.pone.0087366. eCollection 2014. PMID 24520330